CLINICAL TRIAL: NCT05945160
Title: A Randomized Controlled Study Using Alpha Lipoic Acid and CoQ-10 to Determine if Vestibular Function Can be Improved or Maintained Over the Course of One Year
Brief Title: Vestibular Function Using Mitochondrial Antioxidant Therapy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding was terminated, the study will not enroll any subjects
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20230134H; 5P30AG044271 (NIH)
Record Dates: First submitted 2023-07-05; First posted 2023-07-14 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Vestibular Function Disorder
Keywords: Alpha lipoic acid; CoQ10
MeSH Terms: conditions — Vestibular Diseases | interventions — Thioctic Acid; coenzyme Q10

STUDY DESIGN:
Intervention Model Description: Two arm non-blinded controlled clinical trial. Subjects will be randomized 1: 1 either into the investigational antioxidant arm or the standard of care, no study drug arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplements Group (Experimental): Alpha Lipoic Acid will be administered as two 300 mg capsules taken once daily CoQ-10 will be administered as two 200mg capsules daily.
  Interventions: Drug: Alpha Lipoic Acid 300mg; Drug: Coenzyme Q10 200mg
- Standard of Care Group (No Intervention): Standard of care treatment for vestibular function.

INTERVENTIONS:
Drug: Alpha Lipoic Acid 300mg — A naturally occuring mitochondrial antioxidant
  Other Names: ALA
  Arms: Nutritional Supplements Group
Drug: Coenzyme Q10 200mg — A naturally occuring mitochondrial antioxidant
  Other Names: CoQ10
  Arms: Nutritional Supplements Group

SUMMARY:
To determine if supplementation with known mitochondrial antioxidants (alpha lipoic acid (ALA) and CoQ-10) will stabilize or improve vestibular function in older adults.

DETAILED DESCRIPTION:
The subjects will be divided into two groups, half will be given daily supplementation with ALA and CoQ-10. The second group will only receive standard of care treatment, with no study drug intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Community dwelling non-gender specific aged 65-90 years of age
2. For female subjects, confirm that they are post-menopausal
3. Diagnosed with vestibular dysfunction
4. Able to provide informed consent
5. Prepared to adhere to study drug regimen and attend all study visits

Exclusion Criteria:

1. Unable to provide informed consent
2. Allergy/sensitivity to the study drugs or any of their ingredients
3. Unable to adhere to study drug regimen or to attend study visits.
4. Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention.
5. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
6. Anticoagulant drugs: Anisindione (Miradon), dicumarol and warfarin (Coumadin and Jantoven)
7. Participants who are currently undergoing treatment with Insulin, Levothyroxine or chemotherapy drugs.
8. Participants who are undergoing treatment with theophylline.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Slow Harmonic Acceleration | Baseline to 12 months
  Change in vestibular function using the slow harmonic acceleration rotating chair test to measure change, phase and time constant. The sinusoidal harmonic acceleration (SHA) test is a diagnostic procedure used to evaluate the vestibular system, which is responsible for maintaining balance. In the sinusoidal harmonic acceleration test, a person sits in a rotational chair that moves smoothly in controlled, rhythmic oscillations. These movements stimulate the vestibular system and induce eye movements that reflect dynamic vestibular function. Abnormal findings on the SHA test may suggest unilateral or bilateral vestibular dysfunction and provide insights into the status of central compensation for vestibular issues.

SECONDARY OUTCOMES:
Step Velocity Test | Baseline to 12 months
  Step velocity test involves sudden chair rotations and abrupt stops in both directions, which generate compensatory eye movements predominantly in response to the stimulated side. Abnormal findings during this test can suggest problems with the vestibular system, providing additional information about the affected side.
Number of falls | Baseline to 12 months
  A count of number of falls experienced
Tolerance of supplements | Baseline to 12 months
  Number of adverse events experienced

CONTACTS AND LOCATIONS:
Overall Officials: Brian Perry, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study completion when the PI publishes in a peer review journal.